CLINICAL TRIAL: NCT01471600
Title: Randomized Control Study : Safety and Efficacy of Carbohydrate Drink Ingested Two Hours Before Upper Endoscopy Under General Anaesthesia
Brief Title: Safety and Efficacy of Carbohydrate Drink Ingested Two Hours Before Upper Endoscopy Under General Anaesthesia
Acronym: ENDOGLUcide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2008-A00255-50; 08-009 (Other: Caen, Hospital)
Record Dates: First submitted 2011-10-18; First posted 2011-11-15 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Upper Gastrointestinal Endoscopy
Keywords: upper gastrointestinal endoscopy; general anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No intervention (No Intervention): Group overnight fasting
- Group drink (Active Comparator): Glucose drink (200 ml of fruit juice without pulp, ± 200ml coffee or tea, 2 at 4 hours before induction of anaesthesia)
  Interventions: Procedure: group drink

INTERVENTIONS:
Procedure: group drink — group glucose drink : 200 ml of fruit juice without pulp, ± 200ml coffee or tea, 2 at 4 hours before induction of anaesthesia
  Arms: Group drink

SUMMARY:
In several national anaesthesia societies, clear fluids are allowed up to 2 hours before general anaesthesia (GA) and light meals up to 6h. Because of aspiration risk, strict fasting remains routine. Recently, surgical studies proved that pre-operative carbohydrate-rich drink reduces preoperative discomfort without affecting gastric fluid volume and acidity.The aim of this study was to show the effects of preanaesthetic oral fluid in patients undergoing upper endoscopy without emergency. The expected efficacy is a reduction of the preoperative discomfort. The investigators thus propose a randomised prospective open-label study to assess efficacy of preanaesthetic oral glucose drink in patients undergoing upper endoscopy without emergency. Study compare two groups : group "drink" (200 ml of fruit juice without pulp ± 200 ml of coffee or tea, 2 at 4 hours before the induction of anaesthesia) and group "overnight fasting".Discomfort was measured at 2 hours before GA (H-2), just before GA (H0) and 4h after anaesthesia (H+4). Each item (anxiety, thirst, hunger, nervousness, tiredness, nausea) was estimated by visual analogue scale (VAS from 0 to 100mm) and handgrip strength by dynamometer. Gastroenterologist assessed the quality of endoscopy (VAS), gastric residual fluid and acidity.The main aim of this study was to assess in patients referred for upper endoscopy under general anaesthesia, the effect of carbohydrate drink on preanaesthetic discomfort. Secondary purpose were to compare quality of endoscopy, residual gastric volumes, gastric acidity and incidence of side effects. 118 patients will be included in the study. A stratification will be made on the type of endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 yrs
* undergoing upper endoscopy procedure under general anesthesia without emergency
* informed written consent

Exclusion Criteria:

* emergency
* might impair gastrointestinal motility (intestinal obstruction, stenosis)
* diseases of the central and peripheral nervous system or neuromuscular diseases
* drug-induced gastric emptying disorders
* pregnancy
* ionic disorders (hyponatremia<125mmol/l ; hypokalemia<3,5mmol/l
* hemodynamic disorders (systolic arterial pressure <100mmHg)
* unstable diabetes (glycemia>2,5g/l) ± insulin- dependent diabetes ± diabetic gastroparesis
* the potential for difficult airway management
* understanding of the information
* patient with bad prognosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2008-05; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
percentage of preoperative patients increasing the anxiety score just before anaesthesia (H0) | at H0 (just before anaesthesia). The participants will be followed for the duration of hospital stay, an expected average of one day.
  percentage of patients who increased the anxiety score (Visual Analogue Scale of Anxiety) just before anaesthesia.

SECONDARY OUTCOMES:
discomfort (anxiety, thirst, hunger, nervousness, nausea, tiredness) assessed by visual analogue scale (VAS) just before anaesthesia | at H0 (just before anaesthesia). The participants will be followed for the duration of hospital stay, an expected average of one day.
  discomfort (anxiety, thirst, hunger, nervousness, nausea, tiredness) assessed by visual analogue scale (VAS from 0 to 100mmm) just before anaesthesia (at H0).
handgrip strength assessed by dynamometer just before anaesthesia | at H0 (just before anaesthesia). The participants will be followed for the duration of hospital stay, an expected average of one day.
  handgrip strength assessed by dynamometer just before anaesthesia
quality of endoscopy estimated by gastroenterologist by visual analogue scale (VAS from 0 to 100mm) | The participants will be followed for the duration of hospital stay, an expected average of one day.
  quality of endoscopy estimated by gastroenterologist by visual analogue scale (VAS from 0 to 100mm)
gastric residual volume (ml) | The participants will be followed for the duration of hospital stay, an expected average of one day.
  gastric residual volume (ml)
amount of propofol (mg) | The participants will be followed for the duration of hospital stay, an expected average of one day.
  the propofol consumption (mg)
gastric acidity (pH) | The participants will be followed for the duration of hospital stay, an expected average of one day.
  gastric acidity (pH) measured by pH indicator paper
occurrence of vomiting | The participants will be followed for the duration of hospital stay, an expected average of one day.
  occurrence of vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Marie A PIQUET, PhD MD, Principal Investigator — CAEN, Hospital
Locations (1):
- University Hospital, Caen, France